CLINICAL TRIAL: NCT01290861
Title: Cognitive Assessment Battery (CAB)Beta Study
Brief Title: Cognitive Assessment Battery (CAB) Beta Study
Acronym: CAB
Status: Completed | Type: Observational
Sponsor: CHDI Foundation, Inc. (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: CAB Beta
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease; Cognitive Battery; Cognitive Testing; Cognition; pre-manifest Huntington's Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- pre-manifest HD
- early manifest HD
- healthy controls

SUMMARY:
The overall objective of this study is to identify a 60 minute cognitive battery, for subsequent use in clinical trials, that detects cognitive deficits in early HD and late pre-manifest HD compared to controls, and that has a potential to show drug induced improvements.

DETAILED DESCRIPTION:
Huntington's disease (HD) is an autosomal dominant genetic disease which typically manifests beginning in adulthood in the form of movement symptoms, cognitive decline, and psychiatric changes. The proposed research is undertaken in collaboration with CHDI Foundation, Inc., a not for profit organization dedicated to finding treatments for HD. CHDI's goal is to develop or help to develop both symptomatic and disease modifying treatments for HD. To enable future therapeutic trials, CHDI has sponsored several prospective, longitudinal, observational biomarker studies of pre-manifest and early HD with the goal of determining which combination of measures is the most sensitive for detecting changes over the natural progression of pre-manifest and early HD. These and other studies have demonstrated a progressive decline in cognitive function in patients with the huntingtin gene mutation beginning in the pre-manifest period and progressing throughout the course of the disease. These findings support the use of cognitive measures as endpoints in future therapeutic clinical trials. CHDI is committed to the development of a cognitive assessment battery for use in HD therapeutic trials.

There will be paper and pencil and computerized cognitive tests given over a six week period to non-HD control subjects, pre-manifest HD and early manifest HD subjects.

ELIGIBILITY:
Inclusion Criteria:.

1. For early HD group, subjects eligible are persons who meet the following criteria:

   1. Have clinical diagnostic motor features of HD; and
   2. Have huntingtin CAG expansion ≥ 36; and
   3. Have Stage 1 or Stage 2 HD, defined as UHDRS TFC scores between 7 and 13 inclusive.
2. For the late pre-manifest HD group, subjects eligible are persons who meet the following criteria:

   1. Do not have clinical diagnostic motor features of HD; and
   2. Have huntingtin CAG expansion ≥ 39; and
   3. Have Burden of Pathology scores ≥ 300 .
3. For the healthy control group, subjects eligible are persons who meet the following criteria:

   1. Have no known family history of HD; or,
   2. Have known family history of HD but have been tested for the huntingtin CAG expansion and are not at genetic risk for HD (CAG < 36).
4. For all groups, subjects eligible are persons who meet the following criteria:

   1. Are 25 to 55 years of age inclusive;
   2. Education at ISCED level 2 or higher, (see Table 5 below) and no known learning disability affecting reading ability, per investigator assessment and judgement;
   3. Are capable of complying with study procedures, including cognitive testing that requires spoken, written, and computer based responding;
   4. Are ambulatory and do not require skilled nursing care;
   5. Have not had cognitive testing for 2 or more months prior to the participation in cognitive testing for the current study;
   6. Will not have cognitive testing for other purposes during the course of the study; and,
   7. Are capable of providing informed consent.

Education inclusion criterion definition based on ISCED ISCED level 2: Completion of lower secondary general

Australia: Completed junior high school/year 9

Canada: Completed junior high school or junior secondary school or year 9

United Kingdom: Completed Key Stage 3 of secondary school or 'O' levels, or Year 10/Fourth Form (England/Wales); Year 11 (Northern Ireland); 3rd year secondary (Scotland)

United States: Completed junior high school or grade 9

-

Exclusion Criteria:

1. Current use of investigational drugs or participation in a clinical drug trial (unless approved by the CAB Beta study principal investigator or sponsor);
2. Current intoxication, drug or alcohol abuse or dependence (see below for assessment criteria);
3. Unstable or severe psychiatric disorder, including severe depression as indicated by clinician judgment or IDS-SR score ≥ 39;
4. Significant history of or current medical condition with known or confirmed cognitive sequelae, such as moderate to severe traumatic brain injury, multiple sclerosis, etc;
5. Use of psychostimulants (except caffeine) in the 24 hours prior to site visit;
6. Use of benzodiazepines, alcohol, or other sedating drugs in the 12 hours prior to study visit;
7. If using any psychoactive, psychotropic or other medications or nutraceuticals used to treat HD, the use of inappropriate (e.g., non-therapeutically high) or unstable dose over the past 30 days prior to beginning cognitive testing or throughout the study.

Drug and Alcohol Use Assessment

1. In the past six months has your alcohol or drug use caused you to miss work (or your educational obligations, if relevant) or created significant conflicts in your personal relationships?
2. Over the past month, how many days would you estimate you have consumed more than 4 standard drinks per day (3 for women)?
3. Over the past month, how many days would you estimate that you have used recreational drugs?

Exclude patient if:

* #1 = YES or
* #2 + #3= >18 or
* Patient appears intoxicated or if an alcohol odour is detected

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study participants will be pre-HD, early stage HD and control subjects. The cognitive tests will be given to all participants. (only varied by order of administration) in order to determine what measures will be best at detecting cognitive changes associated with HD.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2011-02

CONTACTS AND LOCATIONS:
Overall Officials: Beth Borowsky, Ph.D., Principal Investigator — CHDI Foundation, Inc.; Julie C Stout, Ph.D., Principal Investigator — Monash University
Locations (20):
- United States (12):
  - University of California, San Diego, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of South Florida, Tampa, Florida
  - Rush University, Chicago, Illinois
  - Hereditary Neurological Disease Center, Inc, Wichita, Kansas
  - Albany Medical College, Albany, New York
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
- Australia (2):
  - Monash University/Bethlehem Hospital, Melbourne
  - Westmead Hospital, Sydney
- Center for Movement Disorders, Markham, Ontario, Canada
- United Kingdom (5):
  - Department of Neuropsychiatry, Edgbaston, Birmingham
  - Plymouth Hospitals NHS Trust, Derriford, Plymouth
  - University Hospital of Wales Cardiff, Cardiff, Wales
  - Cambridge Center for Brain Repair, Cambridge
  - University of Manchester, Manchester

REFERENCES:
- See also: Link to funding agency for the CAB Beta study — http://www.highqfoundation.org/